CLINICAL TRIAL: NCT02788669
Title: Prognostic Impact of Immunohistochemical and Molecular Expression of the Endocytosis Receptor LRP1 in Colonic Adenocarcinomas
Brief Title: LRP1 and Colon Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO15124
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-05

CONDITIONS: Colon Cancer; Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Colorectal cancer (CRC) is a major public health problem in France and worldwide. CRC is the third most common cancer in incidence and mortality in France. The vast majority of these cancers are adenocarcinomas that arise sporadically and develop from precursor lesions: adenoma. All CCR with the same disease stage do not have the same prognosis. Various parameters have been identified as factors influencing the prognosis and allows adjustment of the treatment. The poor histoprognostic factors are vessels and nerves invasion by the tumor or the mucinous adenocarcinoma subtype. At the molecular level, the presence of microsatellite instability (MSI) improves the prognosis, while the presence of a BRAF mutation is an independent poor prognostic factor.

LRP-1 is a multifunctional endocytic receptor that belongs to the family of LDL receptors. It is involved in the clearance of matrix proteases. A loss of expression or a decrease of the LRP-1 activity is correlated with an increase of aggressiveness of cancer cells. This effect was demonstrated in vitro in vesicular thyroid carcinomas after LRP-1 blocking. The decrease in the immunohistochemical expression and LRP-1 genomic in hepatocellular carcinomas and lung adenocarcinomas was correlated with a decrease in the overall survival. In CRC, only one immunohistochemical expression study of LRP-1 in colonic adenocarcinoma has been published to date. This study shows that tumor cells express LRP-1, but in nearly half the cases, weaker than in normal colonic cells. The clinical and prognostic impact of LRP-1 expression in colon cancer and its association with a particular molecular or morphological profile has not been studied to date.

In this work, the investigators will study the immunohistochemical and genic expression of LRP-1 in a series of colorectal cancers.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a major public health problem in France and worldwide. CRC is the third most common cancer in incidence and mortality in France. The vast majority of these cancers are adenocarcinomas that arise sporadically and develop from precursor lesions: adenoma. All CRC with the same disease stage do not have the same prognosis. Various parameters have been identified as factors influencing the prognosis and allows adjustment of the treatment. The poor histoprognostic factors are the presence of tumor vessels and nerves invasion or the mucinous adenocarcinoma subtype. At the molecular level, the presence of microsatellite instability (MSI) improves the prognosis, while the presence of a BRAF mutation is an independent poor prognostic factor.

Low density lipoprotein related Protein Receptor 1 (LRP-1) is a multifunctional endocytic receptor that belongs to the family of LDL receptors. He is involved in the clearance of enzymes responsible for the degradation of the extracellular matrix: the matrix proteases. This role of matrix proteolysis modulator associated with a function of cell migration regulator give to this protein an anticancer role. The antitumor property of LRP-1 has been demonstrated in thyroid cancers in vitro. In these studies, loss of LRP-1 expression or a decrease in the LRP-1 activity was correlated with an increase of cancer cells migration and invasion. However, the opposite effect was observed in prostate cancer cell lines.

The clinical impact of the level of LRP-1 expression on overall survival of cancer patients has been assessed in two studies: one on patients suffering from hepatocellular carcinoma and one on patients suffering from primitive lung adenocarcinomas. In both studies, the decrease of immunohistochemical and gene expression of LRP-1 correlated with overall survival decrease. In CRC, only one immunohistochemical expression study of LRP-1 has been published to date. This study shows that adenocarcinomatous cells express LRP-1, but in nearly half the cases, weaker than in normal colonic cells. The clinical and prognostic impact of LRP-1 expression in colon cancer and its association with a particular molecular or morphological profile has not been studied to date.

In this work, the investigators will study the immunohistochemical and genic expression of LRP-1 in a well-characterized series of CRC.

The main objective of this study is to study by genic and immunohistochemical approaches the role of LRP-1 in the aggressiveness of colon adenocarcinomas.

The secondary objective of this study is to search for associations between LRP-1 expression level and morphological or molecular profiles of colonic adenocarcinomas

This study will be the first to explore the expression of LRP-1 in well characterized colon cancers of different morphological and molecular profiles. This study will help to increase knowledge of the prognostic role of LRP-1 in colon cancer and its possible association with clinical, morphological or molecular parameters.

There will be a retrospective cohort study, single center.

The investigators will first design the list of all eligible patients by using a request in the software DIAMIC of th pathology department with component code "colon", damage code "adenocarcinoma " and period "between 2006 and 2012". Patients suffering from Lynch syndrome or other familial cancer syndrome will be excluded of the study. Informed consent will be send to all the selected patients.

Once the patients list will be completed:

* The patients' medical records will be reviewed for: sociodemographic and clinical data colonic tumor location, presence of synchronous metastases, treatment type and duration, patient follow up to the date of 01/06/2014 point (metastases occurrence, disease recurrence, patient death, ...).
* A central review of all pathological slides will be performed for these criteria: adenocarcinoma subtype according to WHO 2010 classification, differentiation, association with polyps and their types, pTNM stage, invasion front and budding, stroma type, presence and amount of tumor necrosis).
* Immunohistochemical analysis on formalin fixed and paraffin embedded tissue will be performed:

  * qualitative and semi-quantitative evaluation of LRP1 immunoexpression with anti-5A6 and 8G1 antibodies
  * RER phenotype research (MLH1, MSH2, MSH6 and PMS2 immunohistochemistry) and BRAF V600E immunohistochemistry
* Molecular analyzes:

  * analysis of LRP-1 gene expression on frozen tissue
  * for selected cases: search for microsatellite instability, search for BRAF V600E, KRAS (exon 2, 3 and 4) and NRAS (exons 2, 3 and 4) mutation on formalin fixed and paraffin embedded tissue

Statistical analysis:

* Data description: mean and standard deviation for quantitative variables; number and percentage for categorical variables.
* Comparison of tumors having a high expression of LRP-1 and tumors not or little expressing LRP-1 by univariate analysis (Student's test and the Wilcoxon test, Chi2 or Fisher's exact) and multivariate (logistic regression).
* Search factors associated with patient outcomes, including the expression of LRP1, by univariate analysis (log-rank test) and multivariate (Cox model).

Colorectal cancer (CRC) is a major public health problem in France and worldwide. CRC is the third most common cancer in incidence and mortality in France. The vast majority of these cancers are adenocarcinomas that arise sporadically and develop from precursor lesions: adenoma. All CRC with the same disease stage do not have the same prognosis. Various parameters have been identified as factors influencing the prognosis and allows adjustment of the treatment. The poor histoprognostic factors are the presence of tumor vessels and nerves invasion or the mucinous adenocarcinoma subtype. At the molecular level, the presence of microsatellite instability (MSI) improves the prognosis, while the presence of a BRAF mutation is an independent poor prognostic factor.

Low density lipoprotein related Protein Receptor 1 (LRP-1) is a multifunctional endocytic receptor that belongs to the family of LDL receptors. He is involved in the clearance of enzymes responsible for the degradation of the extracellular matrix: the matrix proteases. This role of matrix proteolysis modulator associated with a function of cell migration regulator give to this protein an anticancer role. The antitumor property of LRP-1 has been demonstrated in thyroid cancers in vitro. In these studies, loss of LRP-1 expression or a decrease in the LRP-1 activity was correlated with an increase of cancer cells migration and invasion. However, the opposite effect was observed in prostate cancer cell lines.

The clinical impact of the level of LRP-1 expression on overall survival of cancer patients has been assessed in two studies: one on patients suffering from hepatocellular carcinoma and one on patients suffering from primitive lung adenocarcinomas. In both studies, the decrease of immunohistochemical and gene expression of LRP-1 correlated with overall survival decrease. In CRC, only one immunohistochemical expression study of LRP-1 has been published to date. This study shows that adenocarcinomatous cells express LRP-1, but in nearly half the cases, weaker than in normal colonic cells. The clinical and prognostic impact of LRP-1 expression in colon cancer and its association with a particular molecular or morphological profile has not been studied to date.

In this work, the investigators will study the immunohistochemical and genic expression of LRP-1 in a well-characterized series of CRC.

The main objective of this study is to study by genic and immunohistochemical approaches the role of LRP-1 in the aggressiveness of colon adenocarcinomas.

The secondary objective of this study is to search for associations between LRP-1 expression level and morphological or molecular profiles of colonic adenocarcinomas

This study will be the first to explore the expression of LRP-1 in well characterized colon cancers of different morphological and molecular profiles. This study will help to increase knowledge of the prognostic role of LRP-1 in colon cancer and its possible association with clinical, morphological or molecular parameters.

There will be a retrospective cohort study, single center.

The investigators will first design the list of all eligible patients by using a request in the software DIAMIC of th pathology department with component code "colon", damage code "adenocarcinoma " and period "between 2006 and 2012". Patients suffering from Lynch syndrome or other familial cancer syndrome will be excluded of the study. Informed consent will be send to all the selected patients.

Once the patients list will be completed:

* The patients' medical records will be reviewed for: sociodemographic and clinical data colonic tumor location, presence of synchronous metastases, treatment type and duration, patient follow up to the date of 01/06/2014 point (metastases occurrence, disease recurrence, patient death, ...).
* A central review of all pathological slides will be performed for these criteria: adenocarcinoma subtype according to WHO 2010 classification, differentiation, association with polyps and their types, pTNM stage, invasion front and budding, stroma type, presence and amount of tumor necrosis).
* Immunohistochemical analysis on formalin fixed and paraffin embedded tissue will be performed:

  * qualitative and semi-quantitative evaluation of LRP1 immunoexpression with anti-5A6 and 8G1 antibodies
  * RER phenotype research (MLH1, MSH2, MSH6 and PMS2 immunohistochemistry) and BRAF V600E immunohistochemistry
* Molecular analyzes:

  * analysis of LRP-1 gene expression on frozen tissue
  * for selected cases: search for microsatellite instability, search for BRAF V600E, KRAS (exon 2, 3 and 4) and NRAS (exons 2, 3 and 4) mutation on formalin fixed and paraffin embedded tissue

Statistical analysis:

* Data description: mean and standard deviation for quantitative variables; number and percentage for categorical variables.
* Comparison of tumors having a high expression of LRP-1 and tumors not or little expressing LRP-1 by univariate analysis (Student's test and the Wilcoxon test, Chi2 or Fisher's exact) and multivariate (logistic regression).
* Search factors associated with patient outcomes, including the expression of LRP1, by univariate analysis (log-rank test) and multivariate (Cox model).

ELIGIBILITY:
Inclusion Criteria:

* patients operated for colon adenocarcinoma infiltrating stage II at least
* operated at Chu Reims between 01/01/2006 and 31/12/2012
* who have given their consent for this study
* did not receive treatment neoadjuvant.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with sporadic colonic adenocarcinoma treated by surgery at the Academic Hospital of Reims without any neoadjuvant therapy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
LRP1 molecular expression | between 2006 and 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France, France

REFERENCES:
- [Background] Galissier T, Schneider C, Nasri S, Kanagaratnam L, Fichel C, Coquelet C, Diebold MD, Kianmanesh R, Bellon G, Dedieu S, Marchal Bressenot A, Boulagnon-Rombi C. Biobanking of Fresh-Frozen Human Adenocarcinomatous and Normal Colon Tissues: Which Parameters Influence RNA Quality? PLoS One. 2016 Apr 28;11(4):e0154326. doi: 10.1371/journal.pone.0154326. eCollection 2016. PMID 27124490